CLINICAL TRIAL: NCT00813605
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety and Efficacy of FOLFIRI in Combination With AMG 479 or AMG 655 Versus FOLFIRI for the Second-line Treatment of KRAS-mutant Metastatic Colorectal Carcinoma
Brief Title: QUILT-2.018: Safety & Efficacy of FOLFIRI With AMG 479 or AMG 655 vs FOLFIRI Alone in KRAS-mutant Metastatic Colorectal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NantCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20060579; QUILT-2.018 (Other: NantCell, Inc.)
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: AMG 655; AMG 479; Colon Cancer; Rectal Cancer; Monoclonal Antibody; Clinical Trial; Colorectal Cancer; metastatic colorectal cancer; metastatic cancer; antibody-2nd line; KRAS; adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Neoplasm Metastasis; Adenocarcinoma | interventions — IFL protocol; conatumumab; ganitumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental): AMG 655 10 mg/kg plus AMG 479 placebo in combination with FOLFIRI every 14 days
  Interventions: Other: FOLFIRI; Biological: AMG 655; Other: Placebo
- Arm C (Active Comparator): AMG 479 Placebo plus AMG 655 Placebo in combination with FOLFIRI every 14 days
  Interventions: Other: FOLFIRI; Other: Placebo
- Arm B (Experimental): AMG 479 12 mg/kg plus AMG 655 placebo in combination with FOLFIRI every 14 days
  Interventions: Other: FOLFIRI; Other: Placebo; Biological: AMG 479

INTERVENTIONS:
Other: FOLFIRI — Day 1 of each Cycle
  Combination Therapy of:
  irinotecan 180 mg/m2 90-minute infusion leucovorin 400 mg/m2 2 hour infusion 5-FU 400 mg/m2 IV bolus 5-FU 2,400 mg/m2 46-48 hour infusion
Biological: AMG 655 — AMG 655 is an investigational, fully human, monoclonal antibody that selectively binds to Death Receptor-5 (DR-5)
  Other Names: Conatumumab
  Arms: Arm A
Other: Placebo — Inactive dummy agent (to maintain blind)
Biological: AMG 479 — AMG 479 is an investigational, fully human, monoclonal antibody that binds with Insulin-like growth factor receptor type 1
  Arms: Arm B

SUMMARY:
This is a phase 2, multicenter, randomized, double-blind, double-dummy, placebo-controlled, three-arm trial to be conducted in the United States, Europe, and Asia. Approximately 150 eligible KRAS-mutant metastatic colorectal cancer subjects who have failed first line fluoropyrimidine and oxaliplatin-based regimen with or without anti-VEGF therapy will be randomized in a 1:1:1 ratio to receive AMG 479 placebo plus AMG 655 with FOLFIRI, or AMG 479 plus AMG 655 placebo with FOLFIRI, or AMG 479 placebo plus AMG 655 placebo with FOLFIRI

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of colon or rectum in patients with metastatic disease
* Mutant-type KRAS tumor at screening
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 1
* Adequate hematology, renal, hepatic, and coagulation function

Exclusion Criteria:

* History or known presence of central nervous system metastases
* History of other malignancy
* Prior irinotecan-based chemotherapy for advanced/metastatic disease
* Prior death receptor agonists, or other systemic IGF-1R agonists in any setting
* Uncontrolled cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Length of Study

SECONDARY OUTCOMES:
Overall Survival, Objective Response, Duration of Response, Time to Response | Length of Study
Incidence of adverse events | Length of Study
Significant laboratory abnormalities | Length of Study
Incidence of antibody formation | Length of Study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (60):
- United States (26):
  - Research Site, Beverly Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Santa Maria, California
  - Research Site, Denver, Colorado
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Fishers, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Paducah, Kentucky
  - Research Site, Worcester, Massachusetts
  - Research Site, Lebanon, New Hampshire
  - Research Site, Hudson, New York
  - Research Site, New York, New York
  - Research Site, High Point, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Temple, Texas
  - Research Site, Tyler, Texas
  - Research Site, Roanoke, Virginia
- France (4):
  - Research Site, Bordeaux
  - Research Site, Boulogne-Billancourt
  - Research Site, Lille
  - Research Site, Lyon
- Research Site, New Territories, Hong Kong
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Pécs
  - Research Site, Szeged
- India (7):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Nashik, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Kolkata, West Bengal
  - Research Site, Bangalore
- Italy (3):
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Orbassano
- Poland (3):
  - Research Site, Gdansk
  - Research Site, Gliwice
  - Research Site, Opole
- Russia (7):
  - Research Site, Arkhangelsk
  - Research Site, Kursk
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Ufa
- Research Site, Singapore, Singapore
- Spain (4):
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, L'Hospitalet de Llobregat, CataluÃ±a
  - Research Site, Madrid, Madrid
  - Research Site, Pamplona, Navarre

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com